CLINICAL TRIAL: NCT06860594
Title: A Phase I Trial Combining Triapine With Radiation Therapy for Recurrent Glioblastoma or Astrocytoma
Brief Title: Testing the Addition of an Anti-Cancer Drug, Triapine, to the Usual Radiation Therapy for Recurrent Glioblastoma or Astrocytoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2025-01531; NCI-2025-01531 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PHI-151; 10699 (Other: City of Hope Comprehensive Cancer Center LAO); 10699 (Other: CTEP); UM1CA186717 (NIH)
Record Dates: First submitted 2025-03-05; First posted 2025-03-06 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-10

CONDITIONS: Astrocytoma, IDH-Mutant, Grade 2; Recurrent Adult Diffuse Hemispheric Glioma, H3 G34-Mutant; Recurrent Adult Diffuse Midline Glioma, H3 K27-Mutant; Recurrent Astrocytoma, IDH-Mutant; Recurrent Astrocytoma, IDH-Mutant, Grade 3; Recurrent Astrocytoma, IDH-Mutant, Grade 4; Recurrent Glioblastoma, IDH-Wildtype
MeSH Terms: conditions — Astrocytoma; Lymphoma, Follicular; Glioblastoma | interventions — Specimen Handling; Radiotherapy, Intensity-Modulated; Magnetic Resonance Spectroscopy; 3-aminopyridine-2-carboxaldehyde thiosemicarbazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (IMRT, triapine) (Experimental): Patients undergo IMRT QD 5 days per week (Monday-Friday) for a total of 10 treatment days over 2 weeks and receive triapine PO 2 hours prior to IMRT on each radiation treatment day in the absence of disease progression or unacceptable toxicity. Patients also undergo CT and/or MRI throughout the study as well as blood sample collection during screening and on study. Patients may undergo CSF sample collection during screening.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Radiation: Intensity-Modulated Radiation Therapy; Procedure: Magnetic Resonance Imaging; Drug: Triapine

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood and CSF sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Radiation: Intensity-Modulated Radiation Therapy — Undergo IMRT
  Other Names: IMRT; Intensity modulated radiation therapy (procedure); Intensity Modulated RT; Intensity-Modulated Radiotherapy; Radiation, Intensity-Modulated Radiotherapy
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Triapine — Given PO
  Other Names: 3-aminopyridine-2-carboxaldehyde thiosemicarbazone; 3-AP; 3-Apct; OCX-0191; OCX-191; OCX191; PAN-811

SUMMARY:
This phase I trial tests the safety, side effects, and best dose of triapine in combination with radiation therapy in treating patients with glioblastoma or astrocytoma that has come back after a period of improvement (recurrent). Triapine may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Radiation therapy uses high energy x-rays, particles, or radioactive seeds to kill cancer cells and shrink tumors. Giving triapine in combination with radiation therapy may be safe, tolerable, and/or effective in treating patients with recurrent glioblastoma or astrocytoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To identify the safety and maximally tolerated dose (MTD) of oral triapine used in combination with radiation therapy for patients with recurrent glioblastoma (GBM) or astrocytoma.

SECONDARY OBJECTIVES:

I. To observe and record anti-tumor activity. II. To determine the pharmacokinetics of oral triapine in plasma and the central nervous system (CNS).

III. To evaluate the efficacy of triapine when administered in combination with radiation therapy by assessing:

IIIa. Progression-free survival (PFS); IIIb. Overall survival (OS); IIIc. The proportion of patients requiring bevacizumab for symptom control; IIId. The correlation of genetic mutations in select genes (e.g., p53, p16, KRAS, and Pi3k/mTOR/AKT) with tumor response and clinical outcomes.

OUTLINE: This is a dose-escalation study of triapine in combination with radiation therapy.

Patients undergo intensity-modulated radiation therapy (IMRT) once daily (QD) 5 days per week (Monday-Friday) for a total of 10 treatment days over 2 weeks and receive triapine orally (PO) 2 hours prior to IMRT on each radiation treatment day in the absence of disease progression or unacceptable toxicity. Patients also undergo computed tomography (CT) and/or magnetic resonance imaging (MRI) throughout the study as well as blood sample collection during screening and on study. Patients may undergo cerebrospinal fluid (CSF) sample collection during screening.

After completion of study treatment, patients are followed up at 2 weeks after radiation therapy, then every 3 months for up to 5 years from study treatment initiation.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically, molecularly, or cytologically confirmed recurrent astrocytic tumors including:

  * GBM or variants, IDH-wildtype, grade 2-4 (standard curative measures available or not)
  * Astrocytoma, IDH-mutant, grade 2-4 (standard curative measures available or not)
  * Diffuse midline gliomas, including pediatric-type H3 G34 or E3 K27 mutant tumors.
* Tumors ≤ 6 cm in maximal diameter.

  * Patients who had recent resection for recurrent tumor must have measurable disease.
* Patients must have at least a 6-month break from last dose of radiation therapy.

Re-irradiation within 6 months may increase risk for radiation necrosis/edema, which will affect toxicity assessment and patient safety. Additionally, GBM and other high-grade astrocytic tumors can exhibit pseudo-progression within 6 months from completing definitive, 1st line radiation therapy, and re-irradiation during this period will increase risk for misattribution of effect.

* Prior history of standard dose radiation for gliomas of 59.4-60 gray (Gy) in 1.8-2 Gy per fraction (or equivalent or lower) is allowed.
* Patients who received non-standard radiation dose regimen (e.g., 40 Gy, 34-35 Gy, 25 Gy) or stereotactic radiosurgery are eligible as long as there is at least one of the following:

  * A new tumor outside the original radiotherapy field as determined by the investigator.
  * There is histologic confirmation of tumor on biopsy or resection.
  * Imaging findings are consistent with true progressive disease (on standard MRI sequences, MRI spectroscopy/perfusion, or nuclear medicine imaging).
* Age ≥ 18 years. Because no dosing or adverse event data are currently available on the use of triapine in patients < 18 years of age, children are excluded from this study.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 (Karnofsky ≥ 60%).
* Absolute neutrophil count ≥ 1,500/mcL.
* Hemoglobin ≥ 8 g/dL.
* Platelets ≥ 100,000/mcL.
* Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN).
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) ≤ 3 x institutional ULN.
* Creatinine ≤ 1.5 x ULN OR glomerular filtration rate (GFR) ≥ 50 mL/min/1.73 m^2.
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial.
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class II or better.
* Patients must be able to swallow whole capsules.
* Patients must be able to undergo MRIs with contrast. Patients with non-compatible devices with MRI can be eligible if CT scans of sufficient quality are obtained. However, patients without non-compatible devices may not use CT scans to meet this requirement.
* The effects of triapine on the developing human fetus are unknown. For this reason and because ribonucleotide reductase (RNR) inhibitor agent and radiation are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 12 months after finishing study treatment. People of child-bearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [HCG]) within 2 weeks of registration. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 12 months after completion of triapine administration.
* Ability to understand and the willingness to sign a written informed consent document. Legally authorized representatives may sign and give informed consent on behalf of study participants.

Exclusion Criteria:

* Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > grade 1) with the exception of alopecia.
* Patients who are receiving any other investigational agents.
* Patients who are actively taking medications that are known to induce methemoglobinemia (e.g. sulfonamides, nitrofurans, anti-malarials [primaquine, chloroquine], cyclophosphamide, and ifosfamide).
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to triapine.
* Patients with known G6PD deficiency. Testing for G6PD deficiency is not required.
* Patients with uncontrolled intercurrent illness, active infections, or any other significant condition(s) that would make participation in this protocol unreasonably hazardous.
* Pregnant women are excluded from this study because triapine is a RNR inhibitor agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with triapine, breastfeeding should be discontinued if the mother is treated with triapine. These potential risks may also apply to the radiation used in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-07-30 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicity | Up to 28 days
  Will be graded in severity according to the Common Terminology Criteria for Adverse Events version 5.0. Frequency and severity of adverse events and tolerability of the regimen will be collected and summarized with descriptive statistics. The maximum grade for each type of toxicity will be recorded for each patient and frequency tables will be reviewed to determine toxicity patterns. Will employ the Backfill Bayesian Optimal Interval design to guide dose escalation and establish the maximal tolerated dose (MTD). The target toxicity rate for the MTD is = 0.25.

SECONDARY OUTCOMES:
Response rate | Up to 5 years
  Response rate will be categorized based on the Response Assessment in Neuro-Oncology criteria, in which tumor response is based on clinical history, physical exam, and imaging findings. The total number of patients in each response category divided by the total number of evaluable patients determines response rate. An evaluable patient is defined as an eligible patient who received at least one dose of triapine. The response rates will be calculated with corresponding 95% exact Clopper-Pearson confidence intervals.
Plasma pharmacokinetic (PK) parameters | Up to 2 weeks
  Triapine in plasma and peri-tumoral dialysate will be quantified using a validated liquid chromatography-tandem mass spectrometry assay. Plasma PK parameters will be derived and compared to historical controls. Dialysate concentrations will be calculated at multiple time points. Exploratorily, exposure-response relationships will be evaluated.
Progression-free survival | From study enrollment to date of either disease progression or death, assessed up to 5 years
  Will be estimated using Kaplan Meier curves.
Overall survival | From study enrollment to date of death, assessed up to 5 years
  Will be estimated using Kaplan Meier curves.
Proportion of patients who initiated bevacizumab for symptom control | Up to 5 years
  Will be calculated using descriptive statistics.
Tumor tissue biomarkers | Up to 5 years
  The presence of genetic alterations, expression of RRM2, and other molecular gene expression signatures will be descriptive in relation to tumor response and clinical outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie M Yoon, Principal Investigator — City of Hope Comprehensive Cancer Center LAO
Locations (41):
- United States (41):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - UCI Health - Chao Family Comprehensive Cancer Center and Ambulatory Care, Irvine, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Yale University, New Haven, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Coral Springs, Coral Springs, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - UM Sylvester Comprehensive Cancer Center at Doral, Doral, Florida
  - UM Sylvester Comprehensive Cancer Center at Hollywood, Hollywood, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Kendall, Miami, Florida
  - University of Miami Sylvester Comprehensive Cancer Center at Sole Mia, North Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Memorial Hospital East, Shiloh, Illinois
  - University of Kansas Clinical Research Center, Fairway, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - NYU Langone Hospital - Long Island, Mineola, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - University of Wisconsin Carbone Cancer Center - Eastpark Medical Center, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm